CLINICAL TRIAL: NCT06899802
Title: A Two-stage, Randomized, Double-blind, Dose Ranging Phase 2 Trial in Healthy Adult Participants to Investigate Optimal Dose and Dosing Regimen, and to Evaluate Safety and Immunogenicity of the Recombinant MVA-BN-WEV Vaccine
Brief Title: A Phase 2 Trial in Healthy Adult Participants of the Recombinant MVA-BN-WEV Vaccine
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Collaborators: JPM CBRN Medical (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WEV-MVA-002
Record Dates: First submitted 2025-03-06; First posted 2025-03-28 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-07

CONDITIONS: Encephalitis
Keywords: vaccine; equine encephalitis; healthy participants; phase 2
MeSH Terms: conditions — Encephalitis; Encephalomyelitis, Equine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- MVA-BN-WEV Low Dose (Active Comparator): Participants in MVA-BN-WEV Lose Dose group will receive 2 administrations 4 weeks apart with MVA-BN-WEV vaccine of at least MVA-BN-WEV 1.2 x 10E8 Inf.U in Stage 1. 1 additional dose at 1 year after the second administration of the vaccine if Low Dose is the optimal dose for Stage 2.
  Interventions: Biological: MVA-BN-WEV
- MVA-BN-WEV High Dose (Active Comparator): Participants in MVA-BN-WEV High Dose group will receive 2 administrations 4 weeks apart with MVA-BN-WEV vaccine of at least MVA-BN-WEV 3 x 10E8 Inf.U in Stage 1. 1 additional dose at 1 year after the second administration of the vaccine if High Dose is the optimal dose for Stage 2.
  Interventions: Biological: MVA-BN-WEV
- Placebo (Placebo Comparator): Participants in Placebo group will receive 2 administrations 4 weeks apart with Tris-Buffered Saline in Stage 1. 1 additional dose at 1 year after the second administration of Tris-Buffered Saline for Stage 2.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MVA-BN-WEV — MVA-mBN396 (common name MVA-BN-WEV vaccine), is a highly attenuated, live recombinant virus based on the licensed viral vector MVA-BN, provided as a liquid frozen formulation. It is administered as an intramuscular injection.
  Other Names: MVA-mBN396
  Arms: MVA-BN-WEV High Dose; MVA-BN-WEV Low Dose
Other: Placebo — Tris-Buffered Saline (TBS) (placebo) is a clear liquid, free from visible extraneous particles. TBS is acceptable for use as a diluent and for intramuscular injection.
  Other Names: Tris Buffered Saline
  Arms: Placebo

SUMMARY:
This phase 2 clinical trial will investigate an optimal dose, dosing regimen, and evaluate reactogenicity, safety and immunogenicity in healthy adult participants of the recombinant, multivalent MVA-BN-WEV vaccine. MVA-BN-WEV is intended for active immunization for prevention of disease induced by VEEV and EEEV, in persons aged 18 years and older at high risk of exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants ≥18 and ≤50 years of age at screening.
2. General good health, without clinically relevant medical illness, physical exam findings, or laboratory abnormalities, as determined by the investigator.
3. Prior to performance of any trial specific procedures, the participant has read, signed, and dated an informed consent form, having been advised of the risks and benefits of the trial in a language understood by the participant, and has signed the Health Insurance Portability and Accountability Act authorization form.
4. Body mass index (BMI) ≥18.5 and ≤35.

   a. BMI formula for pounds and inches: BMI = (body weight in pounds) × 703 / (body height in inches)m2
5. Female participants should fulfil one of the following criteria:

   1. At least 1 year post-menopausal (amenorrhea > 12 months) at screening.
   2. Surgically sterile (bilateral oophorectomy, bilateral tubal ligation, hysterectomy)
   3. Will use contraceptives as outlined in inclusion criterion 6 from screening until 30 days after last vaccination.
6. Female participants of childbearing potential and male participants who are sexually active with a female partner of childbearing potential must agree to the use of a highly effective method of birth control from at least 30 days prior to administration of the MVA-BN-WEV vaccine to until last vaccination. Note: medically acceptable methods of contraception that may be used by the participant and/or partner include combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomy or abstinence (abstinence only acceptable if refraining from heterosexual intercourse during the entire period of 30 days prior to administration of the MVA BN WEV vaccine until 30 days after last vaccination).
7. Negative human immunodeficiency virus antibody test (anti-HIV), negative hepatitis B surface antigen (HBsAG) and negative antibody to hepatitis C virus.

Exclusion Criteria:

1. Pregnant or breast-feeding women.
2. Participant has an acute or chronic medical condition that, in the opinion of the investigator, would render the trial procedures unsafe or would interfere with the evaluation of the responses, including but not limited to, neurologic, cardiovascular, respiratory, hepatic, hematologic, rheumatologic, endocrine, gastrointestinal, renal, autoimmune, or immunosuppressive conditions.
3. History of or active autoimmune disease; persons with vitiligo or thyroid disease taking thyroid replacement are not excluded.
4. Known or suspected impairment of immunologic functions including, but not limited to, clinically significant liver disease, diabetes mellitus type I, moderate to severe kidney impairment. A known immunodeficiency syndrome.
5. Known or suspected previous alphavirus infections or previous vaccination (EEEV, VEEV, WEEV, Chikungunya).
6. Known or suspected previous smallpox vaccination, vaccination with a poxvirus-based vaccine, or mpox infection.
7. History of malignancy other than squamous cell or basal cell skin cancer, unless there has been surgical excision at least 6 months prior to screening that is considered to have achieved cure. Participants with history of skin cancer must not be vaccinated at the previous tumor site.
8. Clinically significant mental disorder not adequately controlled by medical treatment.
9. Active or recent history of chronic alcohol abuse and/or intravenous and/or nasal drug abuse (within the period of 6 months before screening).
10. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, eg, tris(hydroxymethyl)-amino methane, quail proteins.
11. History of anaphylaxis or severe allergic reaction to any vaccine.
12. Having received any vaccinations or planned vaccinations with a live vaccine within 30 days prior to first or after last trial vaccination.
13. Having received any vaccinations or planned vaccinations with a non-live or ribonucleic acid (RNA-) based vaccine within 14 days prior to first or after each trial vaccination.
14. Recent blood donation (including platelets, plasma, and red blood cells) within 4 weeks prior screening, or planned blood donations during active trial period (ie, until the end of the active trial visit).
15. Chronic systemic administration (defined as more than 14 days) of > 10 mg prednisone (or equivalent)/day or any other immune-modifying drugs during a period starting 3 months prior to administration of the vaccine and ending at the end of the active trial period Visit. The use of topical, inhaled, ophthalmic and nasal glucocorticoids is allowed.
16. Post organ transplant participants whether or not receiving chronic immunosuppressive therapy.
17. Administration or planned administration of immunoglobulins and/or any blood products during a period starting 3 months prior to administration of the vaccine and ending at the end of the active trial period Visit. Receipt of packed red blood cells given for an emergency indication in an otherwise healthy person, and not required as ongoing treatment is not exclusionary (for example packed red blood cells given in emergency during an elective surgery).
18. History of coronary heart disease, myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, uncontrolled high blood pressure, significant arrhythmia with or without corrective/ablative surgery, or any other heart condition under the care of a doctor.
19. Use of any investigational or non-registered drug or vaccine other than the trial vaccine within 30 days preceding the administration of the trial vaccine, or planned administration of such a drug during the trial period until 12 months after the last vaccination visit (stage 1) or 6 months after last vaccination (stage 2).
20. Employment with the investigator or CTS, with direct involvement in the proposed study or other studies under the direction of that investigator or CTS, or relationship to the investigator or CTS employee.
21. Association with Bavarian Nordic as staff, contractors, agents, or business partners or any financial interest in the outcome of the trial.
22. Federal employees and active-duty military personnel.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 411 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Optimal dose of MVA-BN-WEV vaccine in adult participants in terms of immunogenicity based on eastern equine encephalitis virus (EEEV)- and Venezuelan equine encephalitis virus (VEEV)-specific humoral immune responses to the MVA-BN-WEV vaccination. | 2 weeks after second vaccination.
  The participants' serum binding antibody titers of MVA-BN-WEV vaccine as measured by ELISA against EEEV and VEEV at 2 weeks after the second trial vaccination, and the participants' serum neutralizing antibody titers of MVA-BN-WEV vaccine as measured by PRNT against EEEV and VEEV at 2 weeks after the second trial vaccination.
Booster response of MVA-BN-WEV versus placebo in terms of immunogenicity based on EEEV- and VEEV- specific humoral immune responses to the MVA-BN-WEV vaccine. | 2 weeks after third vaccination.
  The participants' serum binding antibody titers of MVA-BN-WEV vaccine as measure by ELISA against EEEV and VEEV at 2 weeks after the third vaccination, and the participants' serum neutralizing antibody titers of MVA-BN-WEV vaccine as measure by PRNT against EEEV and VEEV at 2 weeks after the third vaccination.

SECONDARY OUTCOMES:
Safety and reactogenicity of the MVA-BN-WEV vaccine and placebo in terms of solicited and unsolicited AEs in participants throughout the trial. | Duration of trial (approximately 19 mon) for SAE or AESI or during active trial period (defined as the period from 1st vaccination up to and including the end of active trial period for stage 1 (4 wks after 2nd vaccination)/stage 2 (4 wks after booster).
  Participants reporting:
  Stage 1 and 2:
  * Any SAE, regardless of relationship, throughout the trial (first vaccination through the end of the trial).
  * Any AESI regardless of relationship from first vaccination through the end of the trial.
  Stage 1:
  • Any grade 3 or higher solicited or unsolicited AEs assessed as related to trial vaccine from first vaccination through end of active treatment period stage 1.
  Stage 2:
  • Any grade 3 or higher solicited or unsolicited AEs assessed as related to trial vaccine from third vaccination through end of active treatment period stage 2.
WEEV-specific humoral immune responses to the MVA-BN-WEV vaccine and the VV-specific humoral immune responses to the MVA-BN-WEV vaccine. | 2 weeks after second vaccination.
  * Serum binding antibody titers against WEEV as determined by ELISA, 2 weeks after second vaccination.
  * Seroconversion response in terms of serum binding antibody titers against WEEV, EEEV, and VEEV as determined by ELISA, 2 weeks after second vaccination.
  * Serum neutralizing antibody titers against WEEV, and VV as determined by PRNT, 2 weeks after second vaccination.
  * Seroconversion response in terms of neutralizing antibody titers against WEEV, EEEV, VEEV, and VV as determined by PRNT, 2 weeks after second vaccination.
WEEV-specific humoral immune responses to the MVA-BN-WEV vaccine versus placebo and the VV-specific humoral immune responses to the MVA-BN-WEV vaccine versus placebo. | 2 weeks after third vaccination.
  * Serum binding antibody titers against WEEV as determined by ELISA, 2 weeks after third vaccination.
  * Serum neutralizing antibody titers against WEEV, and VV as determined by PRNT, 2 weeks after third vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A. Fierro, MD, Principal Investigator — Johnson County Clin-Trials
Locations (9):
- United States (9):
  - Benchmark Research, Sacramento, California
  - Lifeline Primary Care, Inc. / CCT Research, Lilburn, Georgia
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Versailles Family Medicine, PLLC/CCT Research, Versailles, Kentucky
  - Benchmark Research, Kenner, Louisiana
  - Jefferson City Medical Group / Avacare, Jefferson City, Missouri
  - Clay-Platte Family Medicine, P.C./CCT Research, Kansas City, Missouri
  - Papillion Research Center/CCT Research, Papillion, Nebraska
  - Benchmark Research, San Angelo, Texas

IPD SHARING:
Plan to Share IPD: No